CLINICAL TRIAL: NCT02023437
Title: A Prospective, Post-Market-Clinical-Follow-Up Study to Investigate the Long-term (3 Months) Safety of Femtosecond-laser Assisted Cataract Surgery
Brief Title: Long-term (3 Months) Safety of Femtosecond-laser Assisted Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1304_3M
Record Dates: First submitted 2013-12-06; First posted 2013-12-30 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Femtosecond laser cataract surgery (Experimental): "Laser group": a pre-fragmentation of the ocular lens will be performed by VICTUS femtosecond laser lens fragmentation procedure.
  Interventions: Device: Femtosecond laser cataract surgery
- Manual cataract surgery (Active Comparator): "Manual": manual group acts as a control group where the lens fragmentation are performed manually without femtosecond laser assisted lens fragmentation
  Interventions: Device: Manual cataract surgery

INTERVENTIONS:
Device: Femtosecond laser cataract surgery — The VICTUS lens fragmentation procedure is part of the femtosecond laser assisted cataract procedure, which generates precise cuts inside the cataractous lens, leading to a softening and fragmentation of the lens.
  Arms: Experimental: Femtosecond laser cataract surgery
Device: Manual cataract surgery — "Manual": manual group acts as a control group where the lens fragmentation are per-formed manually without femtosecond laser assisted lens fragmentation
  Arms: Manual cataract surgery

SUMMARY:
This clinical study is a prospective, post-market-clinical-follow-up study to investigate the long-term (3 months) safety of femtosecond laser assisted cataract surgery as a study follow-up extension to the Study #1304 titled as "A Multi-centre, Multi-surgeon, Randomized, Controlled, Prospective, Post-Market-Clinical-Follow-Up Study to Investigate the Impact of Cataract Grade on the Efficacy and Safety of Femtosecond-laser Assisted Lens Fragmentation Procedure".

ELIGIBILITY:
Only the patients who were successfully enrolled in Study #1304 are eligible for this follow-up extension study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 3 month
  Less or equal adverse events (e.g. retinal detachment, intraocular lens (IOL) malposition, etc.) in "Laser group" (pooled from all cataract grades) compared with "Manual group" (pooled from all cataract grades); p<0.05 will be considered statistically significant. The primary study end point is only based on adverse events and severe adverse events which are related to the treatment procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Stodulka, Dr. Med., Principal Investigator — Gemini clinic, Zlin, Czech Republic 76001; Kasu P Reddy, M.D., Principal Investigator — MaxiVision Laser Centre Private Limited, Hyderabad, India; N Sreelakshmi, M.D., Principal Investigator — MaxiVision Laser Centre Private Limited, Hyderabad, India; Steve Slade, M.D., Study Chair — Slade & Baker Vision Center
Locations (2):
- Gemini Eye Clinic, Zlín, Czechia
- MaxiVision Laser Centre Private Limited, Hyderabad, India